CLINICAL TRIAL: NCT04539457
Title: Managing Appropriate Prescribing in Primary Care COPD Patients With Comorbidities: Evaluation of the Desktop Helper (Number 10) in a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Managing Appropriate Prescribing in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Practitioners Research Institute (Network)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: GPRI19209
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: COPD; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (No Intervention): Neither the 'Desktop Helper (version 10)' will be integrated in the EMR system nor the 'e-learning' will be offered to GPs. However, to prevent attenuation of usual care, GPs will be free to adjust any medication on their own initiative or to use any other aid to decrease inappropriate prescribing in COPD patients.
- Only desktop helper (Active Comparator): Only the 'Desktop Helper (version 10)' will be integrated in the EMR system. Specifically, GPs will receive a notification about the 'Desktop Helper (version 10)'. This notification will inform general practitioners about the option in the Medicom Smart Module to identify COPD patients with comorbidities who have one or more 'medication-comorbidity clashes' (i.e. undesired interactions between medications for COPD and comorbid conditions).
  Interventions: Behavioral: Desktop helper
- Only E-learning (Active Comparator): Only the 'e-learning' will be offered to GPs. Herein, GPs, will be invited to perform an e-learning module which provide information about COPD and their (co)morbidities and the 'medication-comorbidity clashes'.
  Interventions: Behavioral: E-learning
- Both dekstop helper and e-learning (Active Comparator): Both 'Desktop Helper (version 10)' will be implemented in the EMR system. GPs will subsequently be notified about the possibility to detect COPD patients with 'medication-comorbidity clashes'. The implementation of the 'Desktop Helper (version 10), will be accompanied by e-learning offered to GPs. about COPD and their (co)morbidities and the 'medication-comorbidity clashes'.
  Interventions: Behavioral: Desktop helper; Behavioral: E-learning

INTERVENTIONS:
Behavioral: Desktop helper — The 'Desktop Helper (version 10)' is a user-friendly information sheet developed by the IPCRG. This 'Desktop Helper (version 10)' has been developed in co-operation with several clinicians and experts in the field of COPD. These practical guidance and support are a tool for clinicians working in primary care. The 'Desktop Helper (version 10)' contains specific advice to prevent clashes. The specific advice of the 'Desktop Helper (version 10)' will be elaborated in decision trees. These will be integrated and implemented into the MedicomSmart system by Stichting Healthbase. Subsequently, these decision trees will provide GPs to conduct case-finding of COPD patients with 'medication-comorbidity clashes'. These are based on the 'Desktop Helper (version 10)' . Case finding will be done by the GP or the practice nurse (POH).
  Arms: Both dekstop helper and e-learning; Only desktop helper
Behavioral: E-learning — The e-learning module will be explanatory to the 'Desktop Helper (version 10)' how to perform the case-finding and in what way the case-finding can be beneficial to the patients with COPD and their (co)morbidities. This e-learning module will include several example cases and how to deal with the case-finding and the next steps in the process to reduce the (co)morbidity clashes with the medications of COPD. Together with the decision trees as inferred from the 'Desktop Helper (version 10)', the e-learning module is aimed at inducing a behavioral change in prescribing medication to a patient suffering from COPD and one or more (co)morbidities.
  Arms: Both dekstop helper and e-learning; Only E-learning

SUMMARY:
Objective: Reducing inappropriate medications for primary care COPD patients with comorbidities ('medication-comorbidity clashes'), by evaluation of the Desktop Helper (number 10) in a pragmatic cluster randomized controlled trial.

Study design: A four-arm pragmatic cluster randomized controlled trial (cluster RCT), which will be conducted in GP practices in the Netherlands. In the cluster RCT, the control condition (arm 1: care as usual) will be compared with three intervention arms (i.e. arm 2: the 'Desktop Helper (number 10)' , arm 3: an e-learning module, and arm 4: the 'Desktop Helper (number 10)' accompanied by the e-learning module). At baseline and at 26 weeks of follow-up, a data-extraction of comorbidities and prescribed medications will be obtained from the EMR of participating GP practices.

Study population: Primary care patients with COPD who have 1 or more comorbidities and who are prescribed one or more medications.

Intervention (if applicable): Clinical rules to remediate 'medication-comorbidity clashes' as outlined in the 'Desktop Helper (number 10)'. These clinical rules will be implemented in the EMR to enable the identification of patients with 'medication-comorbidity clashes'. In addition, e-learning about these 'medication-comorbidity clashes' will be offered depending on the treatment arm of the trial.

Main study parameters/endpoints: The number of 'medication-comorbidity clashes'.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients with COPD aged 18 years and older with one or more (co)morbidities.
* A clinical GP diagnosis of COPD (ICPC code R95 (emphysema/COPD).
* Presence of one or more of the following (co)morbidities: Glaucoma (ICPC code F93*), Kidney failure / renal insufficiency (ICPC code: U99.01), Tuberculosis (ICPC code: A70, R70), Diabetes (ICPC code: T90, A91.05), Pneumonia (ICPC code: R81, R81.01), Osteoporosis/osteopenia (ICPC code: L95, L95.02, L95.01), Prostate symptoms (ICPC code: Y06, U05.02), Atrium fibrillation (ICPC code: K78, K79, K80, K84.02, K04, K05), Bronchiectasis (ICPC code: R91, R91.02) and Asthma (ICPC code: R96, R96.02)

Exclusion Criteria:

* Have end-stage COPD or a life expectancy < 6 months
* If they underwent a systematic medication review aimed at reducing inappropriate prescribing. Systematic refers to a collaboration with a pharmacist and the adoption of Beers, STOPP and or START criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of COPD patients with one or more 'medication-comorbidity clashes' | 26 weeks
  The primary outcome of the study is the percentage of COPD patients with one or more 'medication-comorbidity clashes' (i.e. undesired interactions between medications for COPD and comorbid conditions).

SECONDARY OUTCOMES:
Percentages of patients with one or more inappropriately prescribed medication | 26 weeks
  This outcome includes:
  * ICS prescription to patients with diabetes, a history of pneumonia, osteoporosis/osteopenia, bronchiectasis, tuberculosis, glaucoma
  * LABA prescription to patients with atrium fibrillation
  * LAMA prescription to patients with chronic kidney disease, prostate symptoms, glaucoma
  * No ICS prescription in patients with asthma

CONTACTS AND LOCATIONS:
Overall Officials: Janwillem Kocks, MD PhD, Principal Investigator — General Practitioners Research Institute
Locations (1):
- General Practitioners Research Institute, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No